CLINICAL TRIAL: NCT03554525
Title: Clinical Trial to Evaluate the Usefulness of the Regular Consumption of a Food Supplement(FAT-BINDER DAMM) on Weight Regain After an Interventional Diet Program on Overweight/Obese People
Brief Title: Weight Regain After Consumption of Food Supplement and Interventional Diet Program
Acronym: fat-binder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4801
Record Dates: First submitted 2018-04-06; First posted 2018-06-13 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Overweight; Weight Loss; Body Weight Changes; Weight Change, Body
Keywords: Obesity; Overweight; Weight Loss; Body weight maintenance; Weight Change, Body; Saccharomyces Cerevisiae; Beta-glucans
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Body Weight Changes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental product : FAT-BINDER DAMM (Experimental): 3 sticks of the dietary supplement (1.4 grams/stick) during 12 months: 2 sticks should be consumed before lunch and 1 stick before dinner.
  Interventions: Dietary Supplement: Fat-binder damm
- Control product : PLACEBO (Placebo Comparator): 3 sticks of the dietary supplement (1.4grams/stick) during 12 months: 2 sticks should be consumed before lunch and 1 stick before dinner.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fat-binder damm — 3 sticks every day during 12 months
  Arms: Experimental product : FAT-BINDER DAMM
Dietary Supplement: Placebo — 3 sticks every day during 12 months
  Arms: Control product : PLACEBO

SUMMARY:
Effect of the dietary supplement (FAT-BINDER DAMM) on weight regain after 9 months of control weight program

DETAILED DESCRIPTION:
* 60 participants will consume experimental product every day 3 sticks of the dietary supplement (1.4 grams/stick) during 12 months: 2 sticks should be consumed before lunch and 1 stick before dinner. During the 12 first weeks, each volunteer will be included on a low weight program (PPP) with an individual hypocaloric diet planning and regular physical adapted activity (PPP period). When PPP period is over, volunteers will continue consuming the product for 9 months more (Post-PPP period).
* 60 participants will consume everyday 3 placebo sticks (1.4 grams/stick) during 12 months: 2 sticks should be consumed before lunch and 1 stick before dinner. During the first 12 weeks, each volunteer will be included on a low weight program (PPP) with an individual hypocaloric diet planning and regular physical adapted activity (PPP period ). When PPP period is over, volunteers will continue consuming the product for 9 months more.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ranging from 18 to 65 years old.
* BMI ≥27 and <40 kg/m2. Overweight type II, obesity type I and II
* Social or familiar environment that prevents from accomplishing the dietary treatment.
* Willingness to follow a balanced hypocaloric diet in order to lose weight and perform regular physical adapted activity.
* Adequate cultural level and understanding of the clinical trial.
* Signed informed consent.

Exclusion Criteria:

* Individuals diagnosed with Diabetes Mellitus type I.
* Individuals diagnosed with Diabetes Mellitus type II on pharmacological treatment.
* Individuals with dyslipidemia on pharmacological treatment.
* Individuals with hypertension on pharmacological treatment uncontrolled.
* Individuals allergic to yeast.
* Individuals with chronic diseases (hepatic, kidney…).
* Individuals who have participated in the last 6 months in a program or clinical trial to lose weight.
* Individuals receiving at least the preceding 2 months a pharmacological treatment that modifies the lipid profile (for example, statins, fibrates, diuretics, corticosteroids, ADOs).
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Weight Regain | 12 months
  Change from baseline in kilograms

SECONDARY OUTCOMES:
Body Mass Index (weight/height^2) | 12 months
  Change from baseline in kg/m^2
Fat mass percentage | 12 months
  Change from baseline in percentage
Body water percentage | 12 months
  Change from baseline in percentage
Lean mass percentage | 12 months
  Change from baseline in percentage
Triglycerides | 12 months
  Change from baseline
Low density lipoprotein cholesterol | 12 months
  Change from baseline
High density lipoprotein cholesterol | 12 months
  Change from baseline
Fiber | 12 months
  Change from baseline
Satiety evaluation | [Just before eating the product; Just after eating; After 60 minutes; After 90 minutes] Fasting for at least 4 hours. Must do it with a snack accompanied and 500 ml water.
  Visual Analog Scale to evaluate motivation-satiety when eating
24 hours Dietary Recall | 12 months
  24 hours Food habits of overweight and obesity people
Sensory perception | Months 6, 7, 8 y 9. Gustatory and olfactory sensory perception of the subjects for the study products.
  Questionnaire of analysis of sensory perception of the food study product. Five questions that are valued on a scale of 0% to 100% asking about the taste and smell of the study product: desire with which the product is taken, taste, smell, consistency and what wait for effectiveness.
International Physical Activity Questionnaire | 12 months
  People physical activity habits

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, PhD, MS, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided